CLINICAL TRIAL: NCT05622422
Title: A Feasibility and Pilot Study of a Person-centered and Strength-based Intervention to Facilitate Patient Empowerment, Patient Activation, Self-management, Health, and Wellness Among Adults With Chronic Disease
Brief Title: A Chronic Disease Self Care Management Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pace University (Other)
Responsible Party: Principal Investigator, Natalie A. Stepanian Ph.D., RN, Assistant Professor, Pace University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1936501-Pace
Record Dates: First submitted 2022-11-14; First posted 2022-11-18 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: mixed method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body Knowleging Program Pilot Study (Experimental): There will be three groups of 10 participants with a chronic disease that will receive the Body knowledging Program. The intervention aims to activate patients' inherent resources and by this, facilitate empowerment, patient activation, and self-care management of their chronic disease. The participants will include people 18 years and older that have been diagnosed with a chronic disease. This pilot study will use a pre-post design. Some of the data will be collected initially, then the intervention will be provided in seven sessions the first three face-to-face at a local community center and then the last four sessions through video conferencing that will be facilitated by three researchers. Data collection will take place at the first session and then again at the seventh session. The participants will be invited back in week nine to attend a video conference focus group to obtain qualitative data. Both qualitative and quantitative data will be analyzed.
  Interventions: Behavioral: EMPOWER-BKP

INTERVENTIONS:
Behavioral: EMPOWER-BKP — The intervention aims to activate patients' inherent resources and by this, facilitate empowerment, patient activation, and self-care management of their chronic disease. The participants will include people 18 years and older that have been diagnosed with a chronic disease. This pilot study will use a pre-post design. Some of the data will be collected initially at the first session and then again at the seventh session. The intervention will be provided in seven sessions the first three will be face-to-face at a community center and then the last four sessions will be through video conferencing and will be facilitated by three researchers. The participants will be invited to a focus group interview in week nine in order to collect quantitative data. Once the sessions are finished both qualitative and quantitative data will be collected and then analyzed.

SUMMARY:
The intervention aims to activate patients' inherent resources and by this, facilitate empowerment, patient activation and self-care management of their chronic disease.

DETAILED DESCRIPTION:
The intervention aims to activate patients' inherent resources and by this, facilitate empowerment, patient activation, and self-care management of their chronic disease. The participants will include people 18 years and older that have been diagnosed with a chronic disease. This pilot study will use a pre-post design. Data will be collected initially and then at the seventh session. The intervention will be provided in seven sessions face-to-face for the first three sessions and then via video conferencing for the last four sessions. Each session is facilitated by three researchers. Once the sessions are finished the participants will be invited to a focus session so that qualitative data can be collected in week nine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

  * Undergoing treatment for chronic illness
  * Cognitive capacity to participate in group formats
  * Able to answer questions from questionnaires
  * Able to read and speak English.
  * Score greater than 18 on the MoCA cognitive test

Exclusion Criteria:

* Major reduction in cognitive capacity (i.e. major strokes, dementia, or other related conditions).
* Serious mental illness that impacts the ability to give consent or limits effective participation within a group discussion as assessed by the PI and RA in consultation following routine study protocols used in the study setting (patients may suffer from mild cognitive impairment but must be able to understand and complete questionnaires and engage in intervention groups).
* Patients in palliative phases of cancer.
* Patients in an acute medical crisis or in need of intensive care. -Patients who attend similar interventions in the same period or within the past 3 months. -

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-22 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The Health Education Impact Questionnaire (heiQ) | 15 minutes
  measures eight self-management skills in people with chronic conditions. Possible scores are on a 4 point likert scale. The scale is 1-4. higher score indicates better self-management, with the exception of the emotional wellbeing construct for which scoring is reversed.
The Brief Illness Perception Questionnaire (B-IPQ) | 5 minutes
  assesses the five cognitive illness representations on a five-point Likert scale. The scale is 0-10. A higher score reflects a more threatening view of the illness.
The Patient Activation Measure (PAM) | 10 minutes
  the measure of a person's knowledge, skills, and confidence to manage their own health and well-being on a 0-100 scale the higher score measures indicate higher patient activation.
The European Quality of Life Questionnaire (EQ5D) | 10 minutes
  measures a person's quality of life on a scale 0-100. The higher the score the higher the quality of life.
The Bodyknowledging Questionnaire (BKQ) | 20 minutes
  measures the phases of the Bodyknowledging program

CONTACTS AND LOCATIONS:
Overall Officials: Natalie A Stepanian, Ph.D., Principal Investigator — Pace University

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared with other researchers.